CLINICAL TRIAL: NCT05578378
Title: Cladribine Combined With G-CSF and Cytarabine as a Salvage Treatment in Refractory/Relapsed Acute Lymphoblastic Leukemia
Brief Title: Cladribine Combined With G-CSF and Cytarabine as a Salvage Treatment in R/R ALL
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: The First People's Hospital of Changzhou (Other); Zhongda Hospital (Other); Suzhou Municipal Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022027
Record Dates: First submitted 2022-10-05; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-01

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cladribine; Granulocyte Colony-Stimulating Factor; Cytarabine; fludarabine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CLAG arm (Experimental): Cladribine (5 mg/m2)should be intravenous use on day 1-5, granulocyte colony-stimulating factor will be hypodermic injection using 300 μg per day on days 0-5,cytarabine (1.5 mg/m2) every 12 hours, intravenous infusion on day1-5,4 weeks per cycle.
  Interventions: Drug: Cladribine
- Control arm (Active Comparator): Patients in the control arm received the investigator's choice of one of the following three regimens:
  1. FLAG:Fludarabine(30mg/m2)should be intravenous use on day 1-5, granulocyte colony-stimulating factor will be hypodermic injection using 300 μg per day on days 0-5,cytarabine (1.5 mg/m2) every 12 hours, intravenous infusion on day1-5,4 weeks per cycle.
  2. a high-dose cytosine arabinoside-based regimen;
  3. a high-dose methotrexate-based regimen
  Interventions: Drug: Fludarabine

INTERVENTIONS:
Drug: Cladribine — Cladribine combine with cytarabine will be intravenous on days 1-5; G-CSF will be hypodermic injection on day0-5,4 weeks per cycle.
  Other Names: G-CSF; Cytarabine
  Arms: CLAG arm
Drug: Fludarabine — Control arm
  Patients in the control arm received the investigator's choice of one of the following three regimens:
  FLAG:Fludarabine(30mg/m2)should be intravenous use on day 1-5, granulocyte colony-stimulating factor will be hypodermic injection using 300 μg per day on days 0-5,cytarabine (1.5 mg/m2) every 12 hours, intravenous infusion on day1-5,4 weeks per cycle.
  a high-dose cytosine arabinoside-based regimen; a high-dose methotrexate-based regimen
  Other Names: cytosine arabinoside; methotrexate
  Arms: Control arm

SUMMARY:
To explore the efficiency and safety of CLAG regimen in R/R ALL

DETAILED DESCRIPTION:
R/R Acute Lymphoblastic Leukemia has poor response to second-line chemotherapy.Here,we want to explore efficiency and safety of CLAG regimen in R/R ALL.

ELIGIBILITY:
Inclusion Criteria:

The patients meet the diagnostic criteria for Relapsed/Refractroy B-ALL. ECOG score is 0-3. Expecting life span is more than 6 weeks.

Exclusion Criteria:

Patients are combined with severe organ dysfunction or organ failure: Cardiac failure, Liver and kidney insufficiency.

Patients are combined with severe infection or other complications that can not tolerate chemotherapy.

Patients are considered as other tumor progression. Patients have used cladribine. Pregnant and lactating women will not be included.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
CR (complete remission rate) | the first cycle (4 weeks)
  Response to CLAG regimen.

SECONDARY OUTCOMES:
Overall survival(OS) | From the 1st day to the 365th day after enrollment.
  The time from randomization to death from any cause.
Progression-Free Survival （PFS） | From the 1st day to the 365th day after enrollment.
  It is defined as the total survival of a patient after CR until the tumor recurrence or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Yue Han, MD/PhD, Principal Investigator — Study Principle investigator
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gokbuget N, Stanze D, Beck J, Diedrich H, Horst HA, Huttmann A, Kobbe G, Kreuzer KA, Leimer L, Reichle A, Schaich M, Schwartz S, Serve H, Starck M, Stelljes M, Stuhlmann R, Viardot A, Wendelin K, Freund M, Hoelzer D; German Multicenter Study Group for Adult Acute Lymphoblastic Leukemia. Outcome of relapsed adult lymphoblastic leukemia depends on response to salvage chemotherapy, prognostic factors, and performance of stem cell transplantation. Blood. 2012 Sep 6;120(10):2032-41. doi: 10.1182/blood-2011-12-399287. Epub 2012 Apr 4. PMID 22493293